CLINICAL TRIAL: NCT01672281
Title: Influence of vibroX-training on the Power-duration-relationship and Maximal Force in Relation to Conventional Resistance Training in Endurance Trained Men
Brief Title: vibroX-training in Endurance Trained Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: vbx
Record Dates: First submitted 2012-05-25; First posted 2012-08-24 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vibrox training (Experimental)
  Interventions: Other: vibrox- vs. resistance training
- resistance training (Experimental)
  Interventions: Other: vibrox- vs. resistance training

INTERVENTIONS:
Other: vibrox- vs. resistance training — Comparison between two exercise interventions
  Other Names: vibrox

SUMMARY:
In endurance sports competitions such as cycling, an athlete's capacity to sustain submaximum power (i.e. endurance capacity) strongly influences overall race performance. Endurance capacity can be increased by both long, continuous endurance exercise at moderate oxygen consumption, and high-intensity (at or above peak oxygen consumption) interval training. However, it has also been shown that resistance exercise, if performed in addition to endurance exercise, can further enhance endurance capacity. The investigators have recently described a novel training method, which is based on combined vibration and resistance training and superimposed vascular occlusion. Based on the investigators previous results showing that this type of training leads to marked increases in endurance capacity in previously untrained young women, the investigators aim at investigating whether the method is also effective in increasing endurance capacity in highly endurance-trained young men, and whether the method leads to bigger improvements relative to resistance exercise alone. Besides the functional outcomes the investigators are also interested in the specificity of the cellular adaptations with respect to the two trainings methods.

ELIGIBILITY:
Inclusion criteria:

* male
* no fever / no common cold at the beginning of the study
* at least 4 endurance training sessions prior to beginning of study
* age 18-35y
* non-smoker
* no cardiological / orthopedic problems
* no pacemaker
* fulfills health questionnaire's requirements

Exclusion criteria: female

* fever / common cold at beginning of study
* untrained condition (less than 4 endurance training sessions prior to the
* beginning of the study)
* age under 18 oder above 35y
* smoker
* cardiovascular or orthopedic problems
* cardiac pacemaker
* does not fulfill health questionnaire's requirements

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Critical Power | 2 month intervention
  The difference in changes in Critical Power [Watts] are compared between the vibrox- and resistance training group. For this purpose, participants complete pre and post training a cycling ramp test and 4 cycling constant load tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hans H. Jung, Professor MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Mueller SM, Aguayo D, Lunardi F, Ruoss S, Boutellier U, Frese S, Petersen JA, Jung HH, Toigo M. High-load resistance exercise with superimposed vibration and vascular occlusion increases critical power, capillaries and lean mass in endurance-trained men. Eur J Appl Physiol. 2014 Jan;114(1):123-33. doi: 10.1007/s00421-013-2752-2. Epub 2013 Oct 24. PMID 24154560